CLINICAL TRIAL: NCT00577330
Title: The Efficacy of Myalgesin™ for the Support of Joint Function in Patients With Osteoarthritis of the Knee - A Prospective Randomized Controlled Study
Brief Title: Efficacy of Myalgesin™ to Support Joint Function in Patients With Knee Osteoarthritis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ProThera, Inc. (Industry)
Responsible Party: Stuart I. Erner, MD, The Capital Region Progressive Medicine & Longevity Practice
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MYG-01-2006; 20052687
Record Dates: First submitted 2007-12-18; First posted 2007-12-20 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Frankincense; cortex Phellodendron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Myalgesin (Experimental): Subjects receive Myalgesin twice daily
  Interventions: Dietary Supplement: Myalgesin™ (celery seed extract, Boswellia serrata extract, Phellodendron extract)
- Acetaminophen (Active Comparator): Subjects receive acetaminophen 1000 mg three times a day
  Interventions: Dietary Supplement: Myalgesin™ (celery seed extract, Boswellia serrata extract, Phellodendron extract)

INTERVENTIONS:
Dietary Supplement: Myalgesin™ (celery seed extract, Boswellia serrata extract, Phellodendron extract) — Twice daily

SUMMARY:
Myalgesin is a botanical preparation consisting of celery seed extract,extract of dried Boswellia serrata, and dried extract of Phellodendron bark. Component of these extracts have been shown to exert anti-inflammatory effects and to inhibit cyclooxygenase and 5-lipooxygenase. The study is based on the hypothesis that oral administrration of this botanical will support joint function in people with osteoarthritis of the knee and improve symptoms and mobility as measured by the Western Ontario and McMaster Universities (WOMAC) Osteoarthritis Index.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 50-years or older.
* Patients with symptomatic osteoarthritis of the knees as defined by the American College of Rheumatology criteria(traditional format).
* At least moderate pain in the knee (rated at 40 or greater by the subject on a visual analogue scale) for most days during the last month.
* Use of analgesic or anti-inflammatory agents for control of pain for at least 1 month.
* Baseline functional capacity class 1 to 3, in which class 1 is complete ability to carry out usual activities without handicap,class 2 is ability to adequately conduct usual activities despite handicap of discomfort or limited mobility of one or more joints,and class 3 is limited ability to carry out usual activities. (American Rheumatism Association functional class)
* Documented radiographic changes of osteoarthritis on a previous knee radiograph (Kellgren-Lawrence grade of 2 or more).

Exclusion Criteria:

* Age <50-years.
* Body mass index (BMI) equal to or greater than 35 kg/m2.
* Baseline functional class 4 with the subject bedridden or confined to wheelchair, largely or wholly incapacitated and capable of little or no self-care. (American Rheumatism Association functional class)
* Inflammatory arthritis, gout, pseudogout, or Paget's disease.
* Presence of chronic pain syndromes, such as fibromyalgia or reflex sympathetic dystrophy, that may interfere with the assessment of joint symptomatology.
* Severe bursitis of the knee.
* History of acute joint trauma within 30 days of study entry.
* Complete loss of articular cartilage.
* History of total knee replacement.
* Intra-articular/intramuscular corticosteroids within 30 days of study entry.
* Intra-articular hyaluronan and hyalans within 30 days of study entry.
* History of gastrointestinal bleeding within 1 year of study entry.
* Active peptic ulcer disease, gastroesophageal reflux disease, or inflammatory bowel disease.
* Gastrointestinal tract ulceration within 30 days of study entry.
* Severe renal dysfunction defined as a serum creatinine greater than 2 mg/dL.
* Clinically significant liver disease including an aspartate aminotransferase or alanine aminotransferase >2 times the upper limit of normal.
* Unwillingness or inability to abstain from ethanol for the study duration.
* Significant bleeding disorder.
* History of gastric or duodenal surgery.
* Warfarin use.
* Sensitivity to acetaminophen or to any of the components of Myalgesin™.
* Pregnancy.
* Any serious medical, social or psychological condition that, in the opinion of the Principal Investigator, would disqualify a subject from participation.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2006-05; Study Completion 2008-01 (Estimated)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities (WOMAC) Osteoarthritis Index | 90 days

SECONDARY OUTCOMES:
Lesquesne Algofunctional Index | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Stuart I Erner, MD, Principal Investigator — Private Practice
Locations (1):
- Stuart I. Erner, MD, Albany, New York, United States